CLINICAL TRIAL: NCT01635972
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Bupropion
Brief Title: Drug Interaction Study of Multiple Doses of Isavuconazole and a Single Dose of Bupropion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0044
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Bupropion; Healthy Volunteers
Keywords: Isavuconazole; Bupropion; Bupropion hydrochloride; Healthy Volunteers; BAL8557; BAL4815; BAL8728
MeSH Terms: interventions — isavuconazole; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and bupropion (Experimental): Bupropion hydrochloride on Days 1 and 15, Isavuconazole three times per day (TID) on Days 8 and 9, and once daily (QD) on Days 10 thru 20.
  Interventions: Drug: Isavuconazole; Drug: bupropion hydrochloride

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
Drug: bupropion hydrochloride — oral

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of a single dose of bupropion.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive
* The subject's clinical laboratory test results at Screening and Day 1 are within normal limits unless the Investigator considers the abnormality to be "not clinically significant." Results for aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin must not be above the normal range
* Subject agrees to sexual abstinence, or is surgically sterile, or is using a medically acceptable double barrier method to prevent pregnancy during the study and for three weeks after the follow up phone call at the end of the study, or, if female, is postmenopausal

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission on Day -1
* The subject has a positive result for hepatitis B surface antigen or hepatitis C antibodies at Screening or is known to be positive for human immunodeficiency virus
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the Investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) in the last 6 months
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medication within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has received an experimental agent within 30 days or 5 half-lives, whichever is longer, prior to Day -1
* The subject has a history of suicidal behavior and/or ongoing suicidal ideation as assessed using C-SSRS (Columbia - Suicide Severity Rating Scale) at Screening or at Clinic Check-In (any response of "yes" to the Suicidal Ideation questions on the C-SSRS)
* The subject has a current or past history of seizure disorder or epilepsy
* The subject has a current or past history of depression, anorexia nervosa or bulimia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for bupropion (in plasma): AUCinf, AUClast, Cmax | Day 1 at pre-dose and 0.5,1,1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 48, 72,and 96 hours post-dose and Day 15 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,10,12,16, 20, 24, 48, 72, 96,120, and 144 hours post-dose
  Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to the last quantifiable concentration (AUClast), and maximum concentration(Cmax)

SECONDARY OUTCOMES:
PK profile for bupropion (in plasma): t1/2, tmax, CL/F, and Vz/F | Day 1 at pre-dose and 0.5,1,1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 48, 72,and 96 hours post-dose and Day 15 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,10,12,16, 20, 24, 48, 72, 96,120, and 144 hours post-dose
  Apparent terminal elimination half-life (t1/2), Time to attain Cmax (tmax), Apparent body clearance after oral dosing (CL/F), and apparent volume of distribution (Vz/F)
PK profile for hydroxybupropion (in plasma): AUCinf, AUClast, Cmax, t1/2, tmax | Day 1 at pre-dose and 0.5,1,1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 48, 72,and 96 hours post-dose and Day 15 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8,10,12,16, 20, 24, 48, 72, 96,120, and 144 hours post-dose
PK profile for Isavuconazole (in plasma): AUCtau, Cmax, and tmax | Days 14 and 15 at pre-dose and 0.5,1,1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 20 hours post-dose
  AUC during time interval between consecutive dosing (AUCtau)
PK Isavuconazole (in plasma): trough concentration (Ctrough) | Pre-dose on Days 10 through 13 and Days 16 through 19 and on Day 20: predose and 24 hours post-dose
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) and vital signs | Days 1 through 27 (± 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Phama Global Development
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States